CLINICAL TRIAL: NCT00232037
Title: Extension Study to Assess the Long-Term Safety of Tegaserod in Women With Symptoms of Dyspepsia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHTF919D2301E1
Record Dates: First submitted 2005-09-08; First posted 2005-10-04 (Estimated); Last update posted 2008-02-01 (Estimated); Status verified 2008-01

CONDITIONS: Dyspepsia
Keywords: Dyspepsia, gastrointestinal, tegaserod
MeSH Terms: conditions — Dyspepsia | interventions — tegaserod

INTERVENTIONS:
Drug: Tegaserod

SUMMARY:
This study is being done to evaluate the long-term safety of tegaserod in women with symptoms of dyspepsia who have completed the core study. Tegaserod will be evaluated at 6 mg twice daily.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 years and older
* Fulfilled eligibility criteria in CHTF919D2301 (double blind study) and successfully completed the double-blind study

Exclusion Criteria:

- Early discontinuation from the double-blind study

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Enrollment: 359
Dates: Start 2004-09; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Long term safety at 6 months.

SECONDARY OUTCOMES:
Long term safety at 1 year.
Quality of life : Nepean Dyspepsia Index, WPAI, patient perception of study medication-dyspepsia questionaire.
Efficacy on satisfactory relief at month 6 and 12.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — East Hanover NJ
Locations (1):
- Novartis, East Hanover, New Jersey, United States